CLINICAL TRIAL: NCT04458155
Title: Sample Comparison With Siemens® Point-of-care Device for Cardiac Troponin I Assay by Using a Heparin Coated Transfer Device vs. Non-heparin Coated Transfer Device at the Emergency Department (Validation Study 2.0)
Brief Title: Li-Hep vs. Non-Li-Hep Coated Transfer Device
Status: Completed | Type: Observational
Sponsor: VieCuri Medical Centre (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Principal Investigator, Braim Rahel, Dr. B.M. Rahel, Principal investigator, Cardiologist, VieCuri Medical Centre
Other Study IDs: Study number 580; METCZ20200008 (Other: Medical ethical committee); NL72445.096.20 (Other: ToetsingOnline ID/CCMO ID)
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Acute Coronary Syndrome; Chest Pain; Myocardial Infarction; Cardiac Ischemia
Keywords: Troponin; Point-of-care; Acute coronary syndrome; Siemens; Chest pain
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Capillary blood, venous blood and blood plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest pain patients: Patients are eligible for participation if they are admitted to:
  * The cardiac emergency department (ED) because of chest pain for ruling out acute coronary syndrome by troponin analysis
  * The Coronary Care Unit (CCU) with a NSTEMI or post-percutaneous coronary intervention (PCI) STEMI.
  Troponin analysis will be performed according to standard protocol. From every included patient two capillary blood samples and an extra venous blood sample will be drawn during regularly ordered blood work to evaluate HS cTnI levels obtained with the POC instrument.
  Interventions: Device: Siemens® Point-of-care high sensitive troponin I analyzer

INTERVENTIONS:
Device: Siemens® Point-of-care high sensitive troponin I analyzer — Point-of-care (POC) high sensitive troponin I (HS cTnI) analysis in whole blood, plasma and capillary whole blood with the Siemens® device.

SUMMARY:
This study is a prospective, diagnostic, cohort study within the standard care of acute coronary syndrome (ACS) patients. It compares the analytical performance of Siemens® point-of-care high sensitive troponin I testing in venous, plasma and capillary sample types. The investigators hypothesize that there is a good correlation between the Siemens® POC HS cTnI assay results for the three sample types and that the bias between different POC sample types reduces from ~10% to ≤ 5% when using heparinized transfer device for the capillary sample.

DETAILED DESCRIPTION:
In September 2019, the validation study 1.0 started, in which the cTnI result of the Siemens POC device on three sample types are compared. Interim analysis of the sample comparison was performed by regression analysis using Passing and Bablock, and calculating the Pearson correlation coefficient.

The Li-hep Plasma vs Li-hep venous blood show a very good correlation of 1.00-1.03 with an R of >0.99, so the results between these sample types can be used interchangeably. For the capillary sample vs the Li-hep sample (both blood and plasma) the slope is 8-12% higher. With a 8-12% higher response, the capillary test results may not be interchangeably used with the other 2 sample types.

It is remarkable that capillary samples give a higher response, since it was anticipated that the result may be slightly lower due to the possible dilution by interstitial fluid. The investigators hypothesize that the presence of the Li-heparin anti-coagulant in the venous draw lead to a slight reduction of the apparent cTnI concentration. By using a heparin coated transfer device for the capillary samples instead of an uncoated transfer device, this hypothesis will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Referred to cardiac ED with chest pain suspected of ACS; inclusion at arrival (T=0) or one hour after arrival (T=1).
* Subacute STEMI or NSTEMI patients admitted at the CCU who have an indication for coronary angiography but do not need rescue/emergency PCI.
* STEMI patients who already underwent rescue/emergency PCI; inclusion post PCI.

Exclusion Criteria:

* Out of hospital cardiac arrest.
* Patients with sudden onset tachycardia and a frequency of 110 bpm or higher (supraventricular or ventricular).
* Patients who are hemodynamically unstable or in which an acute non-coronary diagnosis is suspected, e.g. pulmonary embolism, thoracic aortic dissection etc.
* Patients recently already admitted for the same set of symptoms at a previous healthcare institution before being transferred to the participating clinical site.
* Patients not willing or not able to provide informed consent due to their medical condition as judged by the physician.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients presented at our cardiology ED or coronary care unit (CCU) are eligible for inclusion if they are 18 years or older and suspected of having an ACS based on history, examination, ECG and regular troponin results from the central laboratory.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Sample comparison | 30 days
  The primary objective is to compare the analytical performance of Siemens® point-of-care high sensitive troponin I testing in different sample types by using the coefficient of variation.
  This comparison will comprise Siemens® POC capillary vs. Siemens® POC venipuncture and vs. Siemens® POC plasma (Sample comparison).
  The primary objective will be achieved by taking:
  * Two capillary samples > one sample with a heparin coated transfer device (drawn from a finger of the right hand) and the other one with a non-heparin coated transfer device. (drawn from a finger of the left hand)
  * One extra venous blood sample > for POC venous and POC plasma analysis.
  Trained clinical staff will collect the different samples. All samples will be collected once, at one time point with a maximum of 10 minutes in between.

SECONDARY OUTCOMES:
Bland-Altman method | 30 days
  To compare the analytical performance of Siemens® point-of-care high sensitive troponin I testing in different sample types by using the Bland-Altman method.
Linear regression and Pearson's correlation. | 30 days
  The relationship between POC sample types by linear regression and Pearson's correlation.
Overview baseline characteristics. | 30 days
  To create an overview of baseline characteristics of the population.
Major adverse cardiac event (MACE) | 30 days
  MACE is is defined as a composite of cardiac death and myocardial infarction.
Modified HEART score | 30 days
  To determine the modified HEART score retrospectively based upon POC capillary results in the population.
Modified HEART score comparison | 30 days
  To compare the retrospectively determined modified HEART score based upon POC capillary heparin coated transfer device with the retrospectively determined modified HEART score based upon POC capillary non-heparin coated transfer device.

CONTACTS AND LOCATIONS:
Overall Officials: Braim Rahel, Dr., Principal Investigator — VieCuri Medical Centre
Locations (1):
- Viecuri Medical Center, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided